CLINICAL TRIAL: NCT01560260
Title: A Phase 2 Study of Linsitinib (OSI-906) in Pediatric and Adult Wild Type Gastrointestinal Stromal Tumors
Brief Title: Linsitinib in Treating Patients With Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00708; NCI-2012-00708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000728619; SARC-022; SARC 022; SARC022 (Other: Sarcoma Alliance for Research Through Collaboration); 8945 (Other: CTEP)
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Carney Complex; Chondrosarcoma; Gastrointestinal Stromal Tumor; Paraganglioma
MeSH Terms: conditions — Carney Complex; Chondrosarcoma; Gastrointestinal Stromal Tumors; Paraganglioma | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

ARMS (1):
- Treatment (linsitinib) (Experimental): Patients receive linsitinib 150mg orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Linsitinib; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Linsitinib — Given PO
  Other Names: IGF-1R inhibitor OSI-906; OSI-906; OSI-906AA
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well linsitinib works in treating younger and adult patients with gastrointestinal stromal tumors. Linsitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate to treatment with OSI-906 (linsitinib) 150mg BID in patients with advanced wild-type (WT) gastrointestinal stromal tumor (GIST).

SECONDARY OBJECTIVES:

I. To determine the clinical benefit rate (CBR) (stable disease [SD] >= 9 months, partial response [PR], or complete response [CR]) in patients with advanced WT GIST treated with OSI-906.

II. To determine the response duration, progression free survival (PFS), and overall survival (OS) in patients with advanced WT GIST treated with OSI-906.

III. To determine the tolerability and adverse event profile of OSI-906 in patients with advanced GIST.

IV. To explore patterns of protein expression in serum and tumor tissues as predictors of response and progression-free survival (PFS) in advanced WT GIST treated with OSI-906.

V. To evaluate the metabolic response to OSI-906 using fludeoxyglucose F 18 (FDG)-positron emission tomography (PET).

VI. To determine if tumor metabolic response correlates with anatomic response and clinical benefit.

VII. To measure changes in tumor metabolism by FDG-PET qualitatively and semi-quantitatively with standard uptake value (SUV) and tumor body ratio (TBR) from baseline to first computed tomography (CT)-response evaluation and correlate the findings with size changes as defined by conventional cross-sectional imaging scans.

VIII. To investigate correlations between glucose, insulin, and candidate tumor tissue and blood biomarkers with FDG-PET metabolic response.

OUTLINE:

Patients receive linsitinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, every 12 weeks for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed gastrointestinal stromal tumor (GIST) with confirmed genotype of wild-type in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory
* Patients will be stratified into pediatric and adult cohorts; patients in the pediatric cohort (age at diagnosis =< 18 years OR diagnosis of Carney Triad or Carney-Stratakis Diad (paraganglioma, pulmonary chondroma) must have received at least sunitinib and have had progression on or intolerance to progression on therapy; patients in the adult cohort (age at diagnosis > 18 years AND no diagnosis of diagnosis of Carney Triad or Carney-Stratakis Diad) have had progression on or intolerance to imatinib therapy as documented by treating physician
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients must have measurable disease defined as lesions that can be measured in 2 dimensions by medical imaging techniques such as CT or magnetic resonance imaging (MRI); ascites, pleural fluid, and lesions seen on PET scan only are not considered measurable
* White blood cells count (WBC) >= 2.0 x 10^9/L (being >= 14 days off growth factors) OR
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (being >= 14 days off growth factors)
* Platelet count >= 75 x 10^9/L
* Total bilirubin =< 1.5 times the upper limit of normal for age
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) (serum glutamate pyruvate transaminase [SGPT]/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x the upper limit of normal (ULN) for the reference lab (=< 5 x the ULN for the reference lab in the presence of known hepatic metastasis, adjusted for age)
* Creatinine clearance > 70 ml/min/1.73m^2 or
* Serum creatinine < 1.5 x ULN per age and gender
* QT interval corrected using Frederica formula (QTcF) interval average of < 450 msec at baseline using the Frederica formula (QTcF)
* No concomitant drugs that prolong the QT corrected (QTc) interval
* No significant cardiac disease
* Fasting blood glucose < 150 mg/dL at baseline
* Hemoglobin A1C (HbA1c) < 7% at screening
* Patients or their legal representative must be able to read, understand and provide written informed consent to participate in the trial
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; women of childbearing potential must provide a negative pregnancy test (serum or urine) within 7days prior to registration
* Patients with diabetes mellitus should have controlled disease on oral medications, defined as: no diabetic ketoacidosis (hyperglycemia, ketonuria, pH < 7.3 and bicarbonate < 15mEq/L) at the time of enrollment or within 30 days prior to enrollment and; no change in oral medications greater than 10% within 30 days prior to enrollment
* Patient must be able to swallow to participate in the study
* Signed informed consent

Exclusion Criteria:

* Time elapsed from previous therapy must be >= 3 weeks except for prior tyrosine kinase inhibitor therapy which can be >= 7 days; patients must be recovered from the effects of any prior surgery, radiotherapy or systemic therapy
* Patients who are receiving any other investigational agents or other anti-cancer therapies other than those administered in this study during protocol treatment
* Patients with diabetes mellitus requiring insulin for control of their diabetes
* Patients with a history of liver cirrhosis
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to linsitinib (OSI-906)
* While cytochrome P450 1A2 (CYP1A2) inhibitors/inducers are not specifically excluded, investigators should be aware that linsitinib (OSI 906) exposure may be altered by the concomitant administration of these drugs
* While cytochrome P450 2C9 (CYP2C9) substrates are not specifically excluded, investigators should be aware that levels of drugs metabolized by CYP2C9 may be increased by the concomitant administration of linsitinib (OSI-906); caution should be used when administering CYP2C9 substrates to patients who are on study drug
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine are prohibited; other less potent CYP1A2 inhibitors/inducers are not excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior treatment with another kinase inhibitor targeting insulin-like growth factor 1 receptor (IGF-1R) pathway, including monoclonal antibodies targeting IGF-1R
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with linsitinib (OSI-906)
* Fertile men and women of childbearing potential not employing an effective method of birth control throughout the trial and for 3 months after last study drug administration in both sexes; women of childbearing potential must have a negative pregnancy test (serum or urine) within the 7 days prior to study drug administration

  * NOTE: Women of childbearing potential include both pre-menopausal women and women within the first 2 years of the onset of menopause
  * NOTE: Effective methods of birth control includes: surgically sterile, barrier device (condom, diaphragm), contraceptive coil, abstinence; oral contraceptive pills (OCPs) alone are not considered an effective method
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Use of drugs that have a known risk of causing Torsades de Pointes (TdP) are prohibited within 14 days prior to initiation of linsitinib (OSI-906)
* Patients with a history of solid organ transplant are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, Principal Investigator — Sarcoma Alliance for Research through Collaboration
Locations (8):
- United States (8):
  - Stanford Cancer Institute, Palo Alto, California
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - Sarcoma Alliance for Research Through Collaboration, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Songdej N, von Mehren M. GIST treatment options after tyrosine kinase inhibitors. Curr Treat Options Oncol. 2014 Sep;15(3):493-506. doi: 10.1007/s11864-014-0295-3. PMID 24952730

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Linsitinib): Patients receive linsitinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Linsitinib: Given PO
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Linsitinib)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Linsitinib): Patients receive linsitinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Linsitinib: Given PO
  Pharmacological Study: Correlative studies
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response or Partial Response Using Response Evaluation Criteria in Solid Tumors Guideline Version 1.1
Description: Determine the response rate, Complete Response (CR) or Partial Response (PR), to treatment with linsitinib (OSI-906) in patients with advanced wild-type (WT) gastrointestional stromal tumor (GIST) as determined by RECIST 1.1.
Time Frame: At 6 months
Population: 0 out of 20 patients had a response
Measure: Number; unit: participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Clinical Benefit Rate Defined as Stable Disease (SD) >= 9 Months, Partial Response (PR) or Complete Response (CR)
Description: Prolonged non-progression is of clinical benefit (CR + PR + SD at 9 months).
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Groups:
- Treatment (Linsitinib): Patients receive linsitinib 150mg PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Linsitinib: Given PO
  Pharmacological Study: Correlative studies
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
percentage of participants | 40

3. Secondary Outcome: Overall Survival (OS)
Description: Analyzed using Kaplan-Meier curves for the all treated and per protocol populations.
Time Frame: Estimates at 9 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
percentage of participants | 80

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Analyzed using Kaplan-Meier curves for the all treated and per protocol populations.
Time Frame: Time from date of enrollment to time of progression or death due to any cause, estimates at 9 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
percentage of participants | 52

5. Secondary Outcome: Response Duration
Description: Analyzed using Kaplan-Meier curves for the all treated and per protocol populations.
Time Frame: Up to 37 weeks
Population: No responses were observed.
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Failure-free Survival
Description: Analyzed using Kaplan-Meier curves for the all treated and per protocol populations
Time Frame: Up to 37 weeks
Population: Data was not collected for this outcome measure due to limited activity seen with the study treatment.
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Tolerability and Adverse Event Profile of Linsitinib
Description: To determine the tolerability and adverse event profile of OSI-906 in patients with advanced GIST.
Time Frame: Up to 37 weeks
Population: 285 Adverse Events reported during the study.
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
Number analyzed (Adverse Events) | 285
Adverse Events
  Related to study drug | 101
  Related to study drug Grade 3 or higher: number analyzed (Adverse Events) | 101
  Related to study drug Grade 3 or higher | 2

8. Secondary Outcome: Patterns of Protein Expression in Serum and Tumor Tissues as Predictors of Response and PFS
Description: To explore patterns of protein expression in serum and tumor tissues as predictors of response and progression-free survival in advanced WT GIST treated with OSI-906. All Insulin Growth Factor Receptor (IGFR) and phosphorylated AKT (pAKT) evaluation was performed in a blinded manner. Distribution and intensity of positive tumor cell staining was assessed for these markers. Loss of succinate dehydrogenase complex flavoprotein subunit A (SDHA) protein expression has been correlated with the presence of a mutation in SDHA. Loss of succinate dehydrogenase complex iron sulfur subunit B (SDHB) protein expression occurs from bi-allelic inactivation of any of the succinate dehydrogenase (SDH) subunit genes. Loss of expression of one member of the complex alters the structure or production of SDH proteins such that the complex is no longer able to form. This results in elevated intracellular levels of succinate as well as loss of demethylase activity.
Time Frame: Up to 37 weeks
Population: Depending on the patient samples available, the available samples varied from 17 to 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Participants
  SDHA deficiency | 6
  SDHB deficiency | 15
  High to intermediate paKT stain: number analyzed (Participants) | 14
  High to intermediate paKT stain | 6
  High expression of IGFR: number analyzed (Participants) | 14
  High expression of IGFR | 10
  Intermediate levels of IGFR: number analyzed (Participants) | 14
  Intermediate levels of IGFR | 4

9. Secondary Outcome: Number of Participants With Metabolic Response to Linsitinib Using FDG-PET.
Description: Evaluate the number of participants with metabolic response to OSI-906 using fluorodeoxyglucose positron emission tomography (FDG-PET). Evaluation of metabolic response to linsitinib based on two criteria (EORTC and PERCIST).
Time Frame: Up to 37 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Participants
  Partial metabolic response rate | 2
  Stable disease metabolic response rate | 11

10. Secondary Outcome: Changes in Tumor Metabolism by FDG-PET Qualitatively and Semi-quantitatively With Standard Uptake Value (SUV)
Description: To measure changes in tumor metabolism by FDG-PET qualitatively and semi-quantitatively with SUV from baseline to first CT response evaluation and correlate the findings with size changes as defined by conventional cross-sectional imaging scans.
  SUVmax determined by: SUVmax = [VOI activity (mCi/ml) * body wt (g)]/injected dose (mCi) SUVpeak determined by identifying the hottest cubic centimeter within a VOI centered on the lesion with the highest FDG.
Time Frame: Baseline and 8 weeks
Measure: Mean (Full Range); unit: Standard uptake value (SUV)
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Standard uptake value (SUV)
  SUVmax | 19 [8 to 28]
  SUVpeak | 16 [7 to 31]

11. Secondary Outcome: Correlations Between Glucose, Insulin, Tumor Tissue and Blood Biomarkers With FDG-PET Metabolic Response.
Description: To investigate correlations between glucose, insulin, tumor tissue and blood biomarkers with FDG-PET metabolic response.
Time Frame: Up to 37 weeks
Population: Data was not collected in correlation to FDG-PET response results.
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Time to Progression
Description: Time to progression will be evaluated using cumulative incidence.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 20
months | 9.1 [1.84 to 30.1]

13. Other Pre Specified Outcome: Determine the Number of Participants With Tumor Metabolic Response Correlating With Anatomic Response and Clinical Benefit.
Description: To determine if the number of participants with tumor metabolic response correlates with anatomic response and clinical benefit.
Time Frame: Up to 37 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Linsitinib)
Number analyzed (Participants) | 17
Participants
  Partial metabolic response | 2
  Stable disease metabolic response | 11

ADVERSE EVENTS:
Arm/Group | Treatment (Linsitinib)
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Linsitinib) (N=20)
Abdominal Distension - Grade 3 (Unrelated) (Gastrointestinal disorders) | 1 (1)
Abdominal Pain - Grade 3 (Unrelated) (Gastrointestinal disorders) | 3 (4)
Constipation - Grade 2 (Unrelated) (Gastrointestinal disorders) | 1 (1)
Edema Limbs - Grade 2 (Unlikely Related) (General disorders) | 1 (1)
Gastric Hemorrhage - Grade 3 (Unrelated) (Gastrointestinal disorders) | 1 (1)
Hyperglycemia - Grade 3 (Definitely Related) (Metabolism and nutrition disorders) | 1 (1)
Hypoxia - Grade 3 (Unlikely Related) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung Infection - Grade 3 (Unrelated) (Infections and infestations) | 1 (1)
Intra-abdominal hemorrhage - Grade 3 (Unrelated) (Gastrointestinal disorders) | 1 (1)
Rash maculo-papular - Grade 3 (Unrelated) (Skin and subcutaneous tissue disorders) | 1 (1)
Pancreatitis - Grade 3 (Unlikely Related) (Gastrointestinal disorders) | 1 (2)
Renal Calculi - Grade 3 (Unrelated) (Renal and urinary disorders) | 1 (1)
Pleural Effusion - Grade 2 (Unlikely Related) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Supraventricular Tachycardia - Grade 2 (Unrelated) (Cardiac disorders) | 1 (1)
Thromboembolic event (Grade 2 - Unlikely Related) (Vascular disorders) | 1 (1)
Upper gastrointestinal hemorrhage - Grade 3 (Unlikely Related) (Gastrointestinal disorders) | 1 (2)
Seizure - Grade 2 (Unrelated) (Nervous system disorders) | 1 (1)
Fistula Repair - Grade 3 (Unrelated) (Surgical and medical procedures) | 1 (1)
Upper gastrointestinal hemorrhage - Grade 3 (Unrelated) (Gastrointestinal disorders) | 1 (1)
Abdominal Pain - Grade 3 (Unlikely Related) (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Linsitinib) (N=20)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 8 (10)
Alanine Aminotransferase Increased (Investigations) | 2 (3)
Alkaline Phosphatase Increased (Investigations) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 2 (3)
Aspartate Aminotransferase Increased (Investigations) | 2 (6)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 (1) — Eosinophilia
Blurred Vision (Eye disorders) | 1 (1)
Chills (General disorders) | 3 (4)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Creatinine Increased (Investigations) | 3 (3)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (13)
Dizziness (Nervous system disorders) | 5 (6)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Edema Limbs (General disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Eye Disorders - Other (Eye disorders) | 1 (1) — Macular Degeneration
Fatigue (General disorders) | 15 (22)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu-like Symptoms (General disorders) | 1 (1)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 (1) — Gas Pain
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 (1) — Right Upper Quadrant Discomfort
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 (1) — Pain at Fistula Site
Gastrointestinal Pain (Gastrointestinal disorders) | 2 (2)
General Disorders and Administration Site Conditions - Other (General disorders) | 1 (1) — Pain
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 (1) — Lactate dehydrogenase (LDH) Elevation
Headache (Nervous system disorders) | 2 (2)
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1 (1) — Massive Hepatomegaly
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Investigations - Other (Investigations) | 1 (1) — Bladder/Rectum Pain
Lipase Increased (Investigations) | 1 (7)
Memory Impairment (Nervous system disorders) | 1 (1)
Metabolism and Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1 (1) — Vitamin D Deficiency
Musculoskeletal and Connective Tissue Disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Leg Cramps
Musculoskeletal and Connective Tissue Disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Left Rib Pain
Musculoskeletal and Connective Tissue Disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Left Shoulder Pain
Musculoskeletal and Connective Tissue Disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Bilateral Rib Pain
Musculoskeletal and Connective Tissue Disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle Cramps, Lower Extremity
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (17)
Nervous System Disorders - Other (Nervous system disorders) | 1 (1) — Herpes Zoster (Left Buttock and Posterior Left Thigh)
Nervous System Disorders - Other (Nervous system disorders) | 1 (1) — Dizziness
Pain (General disorders) | 2 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palmar-plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Renal Colic (Renal and urinary disorders) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Decreased breath sounds at the bases of the lungs bilaterally
Respiratory, Thoracic and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Rhinorrhea
Serum Amylase Increased (Investigations) | 1 (4)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Pain (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Brittle Nails
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Dermatitis on Hands
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Rash Maculopapular
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (12)
Weight Loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less